CLINICAL TRIAL: NCT04395326
Title: Monitoring of Metabolic Adverse Events of Second Generation Antipsychotics in a Naive Pediatric Population Followed in Mental Health Outpatient and Inpatient Clinical Settings (MEMAS Prospective Study)
Brief Title: Monitoring of Metabolic Adverse Events of Second Generation Antipsychotics in a Naive Pediatric Population
Acronym: MEMAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Leila Ben Amor, Clinical Professor, St. Justine's Hospital
Other Study IDs: MP-21-2016-1201
Record Dates: First submitted 2020-05-08; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-04

CONDITIONS: Adverse Drug Event
Keywords: metabolic side effects; naïve pediatric population; second generation antipsychotics; predictive factors; monitoring
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 24 months follow-up: Single-group study Patients have been included for up to 4 weeks after the initiation of Second Generation Antipsychotic (SGA) treatment (baseline)
  Patients under 18 years of age, previously naïve of antipsychotics, starting an SGA or who started an SGA treatment for less than 4 weeks, followed longitudinally at one of the selected recruiting centers, regardless of the diagnosis that motivated the prescription. Comedications and combination of APs are allowed, as this is an observational study.
  The exclusion criteria are the following: participants diagnosed before or at the baseline with diabetes, dyslipidemia, high blood pressure, thyroid dysfunction, hepatic disease, a disorder that can lead to hyperprolactinemia or another disorder that may interfere with the development of the side effects studied in this research, participants taking a drug intended to treat one of the conditions mentioned above before starting the SGA treatment, and pregnancy.

SUMMARY:
Introduction: Second Generation Antipsychotics (SGAs) are widely used in the pediatric population. It is currently established that SGAs may induce undesirable metabolic adverse events (AEs) such as weight gain, metabolic changes in blood lipids or glucose with risk of potential cardiovascular morbidity and mortality. The Canadian Alliance for Monitoring Effectiveness and Safety of Antipsychotics in children (CAMESA) has published recommendations for monitoring the metabolic AEs of SGAs in the pediatric population. Factors that may be associated with the onset of SGA's metabolic AEs and long term consequences are less studied in the literature. The objectives of our research are to evaluate some factors that can influence the development of the SGA's metabolic AEs, and to study clinical adherence to CAMESA guidelines.

Methods and analysis: The MEMAS study (Monitoring des Effets Métaboliques des Antipsychotiques de Seconde Génération) design is a multicenter, prospective, longitudinal observational study with repeated measures of metabolic monitoring up to 24 months of follow-up. Two recruiting centers have been selected for patients under 18 years of age, previously naïve of antipsychotics, starting an SGA or who have started an SGA for less than 4 weeks regardless of the diagnosis that motivated the prescription. Assessments are performed at inclusion and during follow-up for anthropometric measures (AM), blood pressure (BP) and blood tests (BT) at baseline and 1, 2, 3, 6, 9, 12 and 24 months of follow-up.

Ethics and dissemination: The study protocol was approved by the Centre Hospitalier Universitaire (CHU) Sainte-Justine's Research Ethics Board (MP-21-2016-1201) in 2016 and obtained institutional suitability for the "Centre Intégré Universitaire de Santé et de Services Sociaux du Nord-de-l'Île-de-Montréal" (CIUSSS NIM) Research Center in May 2018. For all participants, written consent will be obtained from parents/caregivers as well as the participant's assent in order to enable their participation in this research project. The results of this research will be published.

DETAILED DESCRIPTION:
Objectives The primary objective is to study selected factors that can influence the development of the SGA's metabolic AEs such as the main diagnosis for which the SGA is prescribed, comorbidities, type and dose of AP, metabolic family history (siblings, parents, parents' siblings, grandparents) and the patient's characteristics (age, height, ethnicity, weight, puberty status). We hypothesize that factors such as younger age of exposure, SGA type, higher SGA doses, lower BMI, non-white ethnic status, hospitalization status at baseline and longer treatment duration will be associated with greater weight gain and, potentially, more cardio-metabolic complications. The secondary objective is to evaluate the clinical adherence to CAMESA guidelines for monitoring of SGAs metabolic AEs in current practice. We hypothesize that the monitoring rates will be low.

Trial design The MEMAS study design is a multicenter, prospective, longitudinal observational study with repeated measures of metabolic monitoring up to 24 months of follow-up. Two recruiting centers have been selected. Recruitment started in January 2017 at CHU Sainte-Justine Hospital and in May 2018 at CIUSSS NIM including the Rivière-des-Prairies (HSM RDP) and Albert-Prévost Mental Health Hospitals (HSM AP). Patients have been included for up to 4 weeks after the initiation of SGA treatment (baseline). Patients will be assured a safe follow-up on their pharmacotherapy. Adherence to the proposed follow-up calendar by the CAMESA guidelines will allow for the detection and the early management of potential cardiometabolic AEs of SGAs. Assessments are performed at inclusion and during follow-up for anthropometric measures (AM), blood pressure (BP) and blood tests (BT) at baseline and 1, 2, 3, 6, 9, 12 and 24 months of follow-up. Participation in this study does not lead to any additional risk to current medical practices. Study participation will end when the patient reaches the end of their 24-month follow-up or earlier if the SGA treatment is discontinued. The prescription of SGA (including dose adjustments, end of treatment, switches and comedications) by the treating psychiatrist is clinically naturalistic. However, during this study, if measured parameters reach what is considered a critical value, the psychiatrist will be notified by the nurse or a member of the research team so that the patient can be referred to a specialist in order to have the proper intervention recommended by the CAMESA guidelines (Ho et al., 2011; Raffin et al., 2014).

Measures All anticipated measurements during the follow-up are : Demographic and clinical baseline data, Adherence to treatment, Anthropometric measures (AM), Blood pressure, Blood tests, and The "MEMAS questionnaire on lifestyle habits and stages of puberty".

Blood tests are performed on site for patients included at HSM AP or Sainte-Justine Hospital whenever possible. For patients included at HSM RDP, blood samples are performed in a local community service center (CLSC) or elsewhere, depending on available resources.

Data collection process In each recruitment center, nurses monitor the participant's studied variables according to the CAMESA calendar. Data is collected and coded from participant's medical records by a member of the research team. All data is anonymized and preserved in the participant's research file. All of the collected information will be kept confidential unless authorized by the participant or his caregiver or an exception from the law. The computerized data will be kept on a password protected file and the paper questionnaires will be kept in a locked space. The data collected will be kept for seven years after the end of the study. After this period of time, it will be safely deleted or destroyed by shredding. The parameters collected for the metabolic monitoring of each SGA-treated participant during follow-up were based on the recommendations of CAMESA guidelines as well as on other, more recent, clinical landmark studies (Nielsen et al., 2014; Pringsheim et al., 2011; Raffin et al., 2014; Rubin et al., 2015). This clinical research project does not require any further investigation compared to the standards of best practice.

Statistical analysis

1. Number of subjects required A number of 60 participants per recruitment center was calculated, for a total of 120 participants. The sample size has been estimated based on previous studies, with available data for four SGAs (risperidone, aripiprazole, quetiapine, olanzapine) and treatment duration up to 12 months (Correll et al., 2009; Findling et al., 2010; Marcus et al., 2011; Findling et al., 2013; Arango et al., 2014; Ronsley et al., 2015). For the estimation of the sample size, the BMI-z score was chosen as the primary dependent variable which is a good reflection of the metabolic changes related to weight gain. ANOVA one-way test was used with compared groups being olanzapine (O), risperidone (R), quetiapine (Q) and aripiprazole (A) with an expected distribution of subjects per group of 1:3:2:2 respectively, the power of 0.80 and an alpha of 0.05. The means to be compared were calculated using the BMI-z score at different times ((BMI-z 3 months + BMI-z 6 months + BMI-z 12 months) / 3); these means are as follow: 0.90 (O), 0.68 (R), 0.52 (Q) and 0.32 (A), with the standard deviation (SD) between 0.20 and 0.60. In the absence of an established size effect for the BMI-z score change, we varied the effect size (d) between 0.31 and 0.93, which resulted in an estimated sample size between 24 and 120 subjects. The sample size of our study was calculated as follows (Desu & Raghavarao, 1990): a one-way ANOVA study, sample sizes of 15, 45, 30, and 30 are obtained from the 4 groups whose means are to be compared. The total sample of 120 subjects achieves 80% power to detect differences among the means versus the alternative of equal means using an F test with a 0.05 significance level. The size of the variation in the means is represented by their standard deviation which is 0.19. The common standard deviation within a group is assumed to be 0.60. The effect size is 0.31. Participants will be recruited from the outpatient and inpatient mental health settings of CHU Ste-Justine and CIUSSS NIM. Thus, annually, the estimated number of patients newly treated with an SGA at CHU Sainte-Justine is approximately 30-40 at the Child and Adolescent Mental Health Outpatient Clinic, 5-10 at Gilles de la Tourette Syndrome Outpatient Clinic, 20 at Child and Adolescent Psychiatric Inpatient Unit (6-17 year old) and at CIUSSS NIM, 30-40 at the Child and Adolescent Psychiatric Inpatient Units (6-17 year olds) and 40 at the Outpatient Mental Health Clinics. Thus, considering a sample size of 120 subjects, we believe that the clinical reality will allow a realistic enrollment of approximately 60 subjects at CHU Sainte-Justine and 60 subjects at CIUSSS NIM.
2. Scheduled analyzes Some analyzes will be provided. Mean changes in AM (weight, BMI-z score, waist circumference), fasting glucose, lipids, and blood pressure will be calculated over time for each SGA group. The percentage of patients in each group who meet one of the following conditions will be calculated: an increase of at least 0.5 in BMI-z score or of more than 7% in weight from baseline over time; developing obesity, metabolic syndrome, hyperglycemia, type 2 diabetes or insulin resistance over time according to the previously mentioned criteria (Measures paragraph). Comparison of baseline values between groups will be considered; chi-square test will be used for categorical variables while a Mann-Whitney U test will be used for continuous variables. This method accounts for multiple comparisons. Comparison between SGAs use in mono- (single AP) vs poly-therapy (combination of two or more APs) will be done. Descriptive analysis will be performed for the sociodemographic variables using percentages, means, medians, ratios and frequencies. A separated analysis will be conducted for the subgroup of participants who received a pharmacological treatment in order to treat the SGAs' cardiometabolic AEs. Thus, only the data available before this pharmacological treatment will be included in the main analysis. Incidence of the metabolic complications will be calculated as the proportion of new-onset metabolic complications at each time point divided by the number of patients with available data. A separate analysis will evaluate the impact of the pharmacological treatment introduced to treat the SGA's cardiometabolic AEs; comparisons will be done with the remaining participants.

ELIGIBILITY:
Inclusion Criteria:

* patients under 18 years of age,
* previously AP-naifs,
* starting an SGA or who started an SGA for less than 4 weeks,
* followed longitudinally at one of the selected recruiting center,
* regardless of the diagnosis that motivated the prescription of the SGA medication.

Exclusion Criteria:

* diabetes,
* dyslipidemia,
* high blood pressure,
* thyroid dysfunction,
* hepatic disease,
* hyperprolactinemia,
* taking a medication to treat any of the above conditions before starting SGA treatment and pregnancy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Population Followed in Mental Health Outpatient and Inpatient Clinical Settings treated by second generation antipsychotics for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant's demographic informations | At baseline (inclusion)
  Sex, age, ethnic group, socioeconomic status will be collected
Participant's clinical informations | At baseline (inclusion)
  Several participant's clinical informations will be collected : recruitment center, inpatient or outpatient status, main diagnosis (DSM-5), comorbidities, second generation antipsychotic prescribed and its dosage, co-medication type and dosage. In order to create an equivalence between the doses of APs received, a conversion to an equivalent dose of chlorpromazine will be carried out according to published standards (Woods et al., 2003).
Family metabolic informations | At baseline (inclusion)
  Presence or not of obesity, dyslipidemia, diabetes and gestational diabetes, high blood pressure, cardiovascular disease in parents will be asked ; and reported weight (in kilograms) and height (in meters) of the parents will be collected (but not measured).
Evaluation of Adherence to second generation antipsychotic treatment | At baseline (inclusion)
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 1 month of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 2 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 3 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 6 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 9 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 12 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Evaluation of Adherence to second generation antipsychotic treatment | At 24 months of follow-up
  Compliance will be indirectly estimated by the nurse and/or the treating psychiatrist at each measurement time of the CAMESA calendar, according to a voluntary declaration by the participants. The date of renewal of the psychotropic medication will also be verified using the Quebec medical record database ("Dossier Santé Québec (DSQ)") and compared to the patient's declaration. The adherence will therefore be counted as the number of days of missed SGA dose per week or per month.
Assessment of change of Body Mass Index (BMI) at different times of the study | At baseline, at 1, 2, 3, 6, 9, 12 and 24 months of follow-up
  Assessment of weight and height will be taken using the same instruments and according to a standardized technique. Body Mass Index (BMI) will be calculated with the weight (kilograms) divided by the height squared (m2). Then, the BMI is standardized for sex and age according to the growth charts of the Centers for Disease Control (CDC) (Ogden et al., 2002) in order to obtain the BMI-z score. Significant weight gain is defined by a 0.5 increase in BMI-z score. Being overweight is defined by a BMI-z between the 85th and the 95th percentile. Obesity is defined by a BMI-z equal to or greater than the 95th percentile.
Assessment of change of waist circumference at different times of the study | At baseline, at 1, 2, 3, 6, 9, 12 and 24 months of follow-up
  Waist circumference (centimeters) will be taken using the same instruments and according to a standardized technique. The waist circumference percentiles will be calculated according to established Canadian standards for age and sex (Katzmarzyk et al., 2004).
Assessment of change of Blood pressure at different times of the study | At baseline, at 1, 2, 3, 6, 9, 12 and 24 months of follow-up
  Systolic and diastolic pressures will be assessed and considered abnormal when it is equal to or higher than the 90th percentile to follow pediatric standards (Cook et al. 2003; Weiss et al., 2004).
Assessment of change of fasting lipids level at different times of the study | At baseline, at 3, 6, 12 and 24 months of follow-up
  The threshold values (mmol/L) for fasting lipids are those recommended by the National Cholesterol Education Program (NCEP, 1992), grouped into commonly used categories (Cook et al., 2003) : total cholesterol > 5.15; LDL >3.34; non-HDL cholesterol >3.73; HDL >1.04; triglycerides (0-9 years) >1.12; triglycerides >1.46 (10-19 years).
Assessment of change of fasting glucose level at different times of the study | At baseline, at 3, 6, 12 and 24 months of follow-up
  Laboratory testing includes fasting blood sugar. Diabetes will be defined according to the criteria (fasting glucose ≥ 0.7 mmol/L with confirmation by other test) established by the American Diabetes Association (ADA, 2004).
Assessment of change of fasting insulinemia level at different times of the study | At baseline, at 3, 6, 12 and 24 months of follow-up
  Laboratory testing includes fasting insulinemia level. Insulin resistance will be estimated with the Homeostasis Model Assessment Insulin - Resistance Index (HOMA-IR) = [Insulin (µUI/ml) x glucose (mg/dl)/405] (Matthews et al., 1985). The threshold value of 2.28 will define insulin resistance (Tresaco et al., 2005).
Assessment of change of prolactin level at different times of the study | At baseline, at 3, 12 and 24 months of follow-up
  Laboratory testing includes prolactin level with normal range between 5 to 20 ng/mL.
Assessment of change of thyroid stimulating hormone (TSH) level at different times of the study | At baseline, at 6, 12 and 24 months of follow-up.
  Laboratory testing includes thyroid stimulating hormone level with normal rate < 10 milliunits per liter (mU/L).
Assessment of change of alanine aminotransferase (ALT) level at different times of the study | At baseline, at 6, 12 and 24 months of follow-up
  Laboratory testing includes alanine aminotransferase level with normal range between 5 to 40 U/L.
Assessment of change in responses to the physical activity MEMAS questionnaire at different times of the study | At baseline, at 1, 3, 6, 12 and 24 months of follow-up
  This self-questionnaire using a compilation of different validated items obtained from the United States Youth Risk Behavior Surveillance System (Brener et al, 2013), from Patient-centered Assessment and Counseling for Exercise + Nutrition, a 2-item validated questionnaire for adolescent physical activity (Hardie Murphy et al, 2015; Prochaska et al, 2001) and also include questions on the perception of self-efficacy during exercise (Motl et al, 2000). Screen time questions collect the number of hours spent during weekdays/ends (Schmitz et al, 2004). Items about transportation to school were adapted from the questionnaire of the Canadian branch of the Health Behavior in School-aged Children (Currie et al, 2010; Gropp et al, 2013). Time spent outdoors outside of school hours is evaluated by the International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE)(LeBlanc et al, 2015; Katzmarzyk et al,2013), items are rated from 0 (strongly disagree) to 4 (very much agree).
Assessment of change in responses to the sleep MEMAS questionnaire at different times of the study | At baseline, at 1, 3, 6, 12 and 24 months of follow-up
  This part of the questionnaire compiles items on the duration (in number of hours) and quality of sleep (from " very good " =1 to " very bad " =4). Items were included since the literature seems to point out a link between lack of sleep and obesity (Chaput & Tremblay, 2012; Chen et al., 2008; Fatima et al., 2015; Patel & Hu, 2008).
Assessment of change in responses to the eating habits MEMAS questionnaire at different times of the study | At baseline, at 1, 3, 6, 12 and 24 months of follow-up
  Eating habits will be assessed using a Food Frequency Questionnaire from the Canadian branch of the Health Behavior in School-aged Children study (Currie et al., 2010; Vereecken & Maes, 2003) and culturally adapted by the ISCOLE team. These items are rated from 1 (no day a week) to 6 (5 days a week).
  Additional items concerning snacks while watching television (Van den Bulck & Van Mierlo, 2004), school meals (Johnson et al., 2014), meals from outside. These items are rated from 1 (no day a week) to 6 (5 days a week). Emotional hunger (Striegel-Moore et al., 1999) are also included. These items are rated from 1 (" never or almost never ") to 3 (" usually or always ").
Assessment of change of Tanner scores at different times of the study | At baseline, at 1, 3, 6, 12 and 24 months of follow-up
  Puberty status will be assessed using a questionnaire developed by Morris and Udry (1980) which includes illustrations of the five Tanner stages of pubertal development, accompanied by brief descriptions (stage 1 = no puberty, stade 2 = completed puberty).

CONTACTS AND LOCATIONS:
Overall Officials: Leila Ben Amor, MD, MSc, Study Chair — Sainte Justine Hospital; Drigissa Ilies, MD, MSC, Principal Investigator — Rivières des Praires Hospital
Locations (1):
- Ben Amor Leila, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will be probably able to share some Individual Participant Data but we will need to make a plan for that and to have an agreement from our ethic research comity

REFERENCES:
- [Background] American Diabetes Association; American Psychiatric Association; American Association of Clinical Endocrinologists; North American Association for the Study of Obesity. Consensus development conference on antipsychotic drugs and obesity and diabetes. Diabetes Care. 2004 Feb;27(2):596-601. doi: 10.2337/diacare.27.2.596. No abstract available. PMID 14747245
- [Background] Arango C, Giraldez M, Merchan-Naranjo J, Baeza I, Castro-Fornieles J, Alda JA, Martinez-Cantarero C, Moreno C, de Andres P, Cuerda C, de la Serna E, Correll CU, Fraguas D, Parellada M. Second-generation antipsychotic use in children and adolescents: a six-month prospective cohort study in drug-naive patients. J Am Acad Child Adolesc Psychiatry. 2014 Nov;53(11):1179-90,1190.e1-4. doi: 10.1016/j.jaac.2014.08.009. Epub 2014 Sep 2. PMID 25440308
- [Background] Centers for Disease Control and Prevention (CDC); Brener ND, Kann L, Shanklin S, Kinchen S, Eaton DK, Hawkins J, Flint KH; Centers for Disease Control and Prevention (CDC). Methodology of the Youth Risk Behavior Surveillance System--2013. MMWR Recomm Rep. 2013 Mar 1;62(RR-1):1-20. PMID 23446553
- [Background] Chaput J-P, Tremblay A. Insufficient Sleep as a Contributor to Weight Gain: An Update. Current Obesity Reports. 2012;1(4):245-56.
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] Correll CU, Rummel-Kluge C, Corves C, Kane JM, Leucht S. Antipsychotic combinations vs monotherapy in schizophrenia: a meta-analysis of randomized controlled trials. Schizophr Bull. 2009 Mar;35(2):443-57. doi: 10.1093/schbul/sbn018. Epub 2008 Apr 15. PMID 18417466
- [Background] Dekelbab BH, Abou Ouf HA, Jain I. Prevalence of elevated thyroid-stimulating hormone levels in obese children and adolescents. Endocr Pract. 2010 Mar-Apr;16(2):187-90. doi: 10.4158/EP09176.OR. PMID 19833586
- [Background] Desu M and Raghavarao D. 1990. Sample Size Methodology. Academic Press. New York.
- [Background] Findling RL, Correll CU, Nyilas M, Forbes RA, McQuade RD, Jin N, Ivanova S, Mankoski R, Carson WH, Carlson GA. Aripiprazole for the treatment of pediatric bipolar I disorder: a 30-week, randomized, placebo-controlled study. Bipolar Disord. 2013 Mar;15(2):138-49. doi: 10.1111/bdi.12042. PMID 23437959
- [Background] Findling RL, Johnson JL, McClellan J, Frazier JA, Vitiello B, Hamer RM, Lieberman JA, Ritz L, McNamara NK, Lingler J, Hlastala S, Pierson L, Puglia M, Maloney AE, Kaufman EM, Noyes N, Sikich L. Double-blind maintenance safety and effectiveness findings from the Treatment of Early-Onset Schizophrenia Spectrum (TEOSS) study. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):583-94; quiz 632. doi: 10.1016/j.jaac.2010.03.013. Epub 2010 May 1. PMID 20494268
- [Background] Ho J, Panagiotopoulos C, McCrindle B, Grisaru S, Pringsheim T; Canadian Alliance for Monitoring Effectiveness and Safety of Antipsychotics in Children (CAMESA) guideline group. Management recommendations for metabolic complications associated with second-generation antipsychotic use in children and youth. Paediatr Child Health. 2011 Nov;16(9):575-80. PMID 23115501
- [Background] Katzmarzyk PT. Waist circumference percentiles for Canadian youth 11-18y of age. Eur J Clin Nutr. 2004 Jul;58(7):1011-5. doi: 10.1038/sj.ejcn.1601924. PMID 15220942
- [Background] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS. The International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE): design and methods. BMC Public Health. 2013 Sep 30;13:900. doi: 10.1186/1471-2458-13-900. PMID 24079373
- [Background] Marcus RN, Owen R, Manos G, Mankoski R, Kamen L, McQuade RD, Carson WH, Findling RL. Safety and tolerability of aripiprazole for irritability in pediatric patients with autistic disorder: a 52-week, open-label, multicenter study. J Clin Psychiatry. 2011 Sep;72(9):1270-6. doi: 10.4088/JCP.09m05933. Epub 2011 Jul 26. PMID 21813076
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] National Cholesterol Education Program (NCEP): highlights of the report of the Expert Panel on Blood Cholesterol Levels in Children and Adolescents. Pediatrics. 1992 Mar;89(3):495-501. No abstract available. PMID 1741227
- [Background] Nielsen RE, Laursen MF, Vernal DL, Bisgaard C, Jakobsen H, Steinhausen HC, Correll CU. Risk of diabetes in children and adolescents exposed to antipsychotics: a nationwide 12-year case-control study. J Am Acad Child Adolesc Psychiatry. 2014 Sep;53(9):971-979.e6. doi: 10.1016/j.jaac.2014.04.023. Epub 2014 Jun 23. PMID 25151420
- [Background] Ogden CL, Kuczmarski RJ, Flegal KM, Mei Z, Guo S, Wei R, Grummer-Strawn LM, Curtin LR, Roche AF, Johnson CL. Centers for Disease Control and Prevention 2000 growth charts for the United States: improvements to the 1977 National Center for Health Statistics version. Pediatrics. 2002 Jan;109(1):45-60. doi: 10.1542/peds.109.1.45. PMID 11773541
- [Background] Pringsheim T, Panagiotopoulos C, Davidson J, Ho J; Canadian Alliance for Monitoring Effectiveness and Safety of Antipsychotics in Children (CAMESA) guideline group. Evidence-based recommendations for monitoring safety of second-generation antipsychotics in children and youth. Paediatr Child Health. 2011 Nov;16(9):581-9. PMID 23115502
- [Background] Raffin M, Consoli A, Giannitelli M, Philippe A, Keren B, Bodeau N, Levinson DF, Cohen D, Laurent-Levinson C. Catatonia in Children and Adolescents: A High Rate of Genetic Conditions. J Am Acad Child Adolesc Psychiatry. 2018 Jul;57(7):518-525.e1. doi: 10.1016/j.jaac.2018.03.020. PMID 29960699
- [Background] Ronsley R, Nguyen D, Davidson J, Panagiotopoulos C. Increased Risk of Obesity and Metabolic Dysregulation Following 12 Months of Second-Generation Antipsychotic Treatment in Children: A Prospective Cohort Study. Can J Psychiatry. 2015 Oct;60(10):441-50. doi: 10.1177/070674371506001005. PMID 26720191
- [Background] Rubin DM, Kreider AR, Matone M, Huang YS, Feudtner C, Ross ME, Localio AR. Risk for incident diabetes mellitus following initiation of second-generation antipsychotics among Medicaid-enrolled youths. JAMA Pediatr. 2015 Apr;169(4):e150285. doi: 10.1001/jamapediatrics.2015.0285. Epub 2015 Apr 6. PMID 25844991
- [Background] Tresaco B, Bueno G, Pineda I, Moreno LA, Garagorri JM, Bueno M. Homeostatic model assessment (HOMA) index cut-off values to identify the metabolic syndrome in children. J Physiol Biochem. 2005 Jun;61(2):381-8. doi: 10.1007/BF03167055. PMID 16180336
- [Background] Weiss R, Dziura J, Burgert TS, Tamborlane WV, Taksali SE, Yeckel CW, Allen K, Lopes M, Savoye M, Morrison J, Sherwin RS, Caprio S. Obesity and the metabolic syndrome in children and adolescents. N Engl J Med. 2004 Jun 3;350(23):2362-74. doi: 10.1056/NEJMoa031049. PMID 15175438
- [Background] Woods SW. Chlorpromazine equivalent doses for the newer atypical antipsychotics. J Clin Psychiatry. 2003 Jun;64(6):663-7. doi: 10.4088/jcp.v64n0607. PMID 12823080
- [Background] Zimmet P, Alberti KG, Kaufman F, Tajima N, Silink M, Arslanian S, Wong G, Bennett P, Shaw J, Caprio S; IDF Consensus Group. The metabolic syndrome in children and adolescents - an IDF consensus report. Pediatr Diabetes. 2007 Oct;8(5):299-306. doi: 10.1111/j.1399-5448.2007.00271.x. No abstract available. PMID 17850473
- [Background] Brener ND, Kann L, Kinchen SA, Grunbaum JA, Whalen L, Eaton D, Hawkins J, Ross JG. Methodology of the youth risk behavior surveillance system. MMWR Recomm Rep. 2004 Sep 24;53(RR-12):1-13. PMID 15385915
- [Background] Hardie Murphy M, Rowe DA, Belton S, Woods CB. Validity of a two-item physical activity questionnaire for assessing attainment of physical activity guidelines in youth. BMC Public Health. 2015 Oct 23;15:1080. doi: 10.1186/s12889-015-2418-6. PMID 26498827
- [Background] Prochaska JJ, Sallis JF, Long B. A physical activity screening measure for use with adolescents in primary care. Arch Pediatr Adolesc Med. 2001 May;155(5):554-9. doi: 10.1001/archpedi.155.5.554. PMID 11343497
- [Background] Motl RW, Dishman RK, Trost SG, Saunders RP, Dowda M, Felton G, Ward DS, Pate RR. Factorial validity and invariance of questionnaires measuring social-cognitive determinants of physical activity among adolescent girls. Prev Med. 2000 Nov;31(5):584-94. doi: 10.1006/pmed.2000.0735. PMID 11071840
- [Background] Schmitz KH, Harnack L, Fulton JE, Jacobs DR Jr, Gao S, Lytle LA, Van Coevering P. Reliability and validity of a brief questionnaire to assess television viewing and computer use by middle school children. J Sch Health. 2004 Nov;74(9):370-7. doi: 10.1111/j.1746-1561.2004.tb06632.x. PMID 15656264
- [Background] Currie C, Griebler R, Inchley J, Theunissen A, Molcho M, Samdal O, Dür W. 2010. Health Behaviour in School-aged Children (HBSC) study protocol : Background, methodology and mandatory items for the 2009/10 survey. Edinburgh : CAHRU & Vienna : LBIHPR.
- [Background] Gropp K, Janssen I, Pickett W. Active transportation to school in Canadian youth: should injury be a concern? Inj Prev. 2013 Feb;19(1):64-7. doi: 10.1136/injuryprev-2012-040335. Epub 2012 May 24. PMID 22627782
- [Background] LeBlanc AG, Broyles ST, Chaput JP, Leduc G, Boyer C, Borghese MM, Tremblay MS. Correlates of objectively measured sedentary time and self-reported screen time in Canadian children. Int J Behav Nutr Phys Act. 2015 Mar 18;12:38. doi: 10.1186/s12966-015-0197-1. PMID 25889903
- [Background] Chen X, Beydoun MA, Wang Y. Is sleep duration associated with childhood obesity? A systematic review and meta-analysis. Obesity (Silver Spring). 2008 Feb;16(2):265-74. doi: 10.1038/oby.2007.63. No abstract available. PMID 18239632
- [Background] Fatima Y, Doi SA, Mamun AA. Longitudinal impact of sleep on overweight and obesity in children and adolescents: a systematic review and bias-adjusted meta-analysis. Obes Rev. 2015 Feb;16(2):137-49. doi: 10.1111/obr.12245. Epub 2015 Jan 14. PMID 25589359
- [Background] Patel SR, Hu FB. Short sleep duration and weight gain: a systematic review. Obesity (Silver Spring). 2008 Mar;16(3):643-53. doi: 10.1038/oby.2007.118. Epub 2008 Jan 17. PMID 18239586
- [Background] Vereecken CA, Maes L. A Belgian study on the reliability and relative validity of the Health Behaviour in School-Aged Children food-frequency questionnaire. Public Health Nutr. 2003 Sep;6(6):581-8. doi: 10.1079/phn2003466. PMID 14690039
- [Background] Johnson CL, Dohrmann SM, Kerckove Vd, Diallo MS, Clark J, Mohadjer LK, Burt VL. National Health and Nutrition Examination Survey: National Youth Fitness Survey Estimation Procedures, 2012. Vital Health Stat 2. 2014 Nov;(168):1-25. PMID 25569584
- [Background] Van den Bulck J, Van Mierlo J. Energy intake associated with television viewing in adolescents, a cross sectional study. Appetite. 2004 Oct;43(2):181-4. doi: 10.1016/j.appet.2004.04.007. PMID 15458804
- [Background] Striegel-Moore RH, Morrison JA, Schreiber G, Schumann BC, Crawford PB, Obarzanek E. Emotion-induced eating and sucrose intake in children: the NHLBI Growth and Health Study. Int J Eat Disord. 1999 May;25(4):389-98. doi: 10.1002/(sici)1098-108x(199905)25:43.0.co;2-4. PMID 10202649
- [Background] Morris NM, Udry JR. Validation of a self-administered instrument to assess stage of adolescent development. J Youth Adolesc. 1980 Jun;9(3):271-80. doi: 10.1007/BF02088471. PMID 24318082
- [Derived] Menard ML, Ilies D, Abadie P, Jean-Baptiste T, Choquette R, Huet AS, Ben Amor L. Monitoring of metabolic adverse events of second-generation antipsychotics in a naive paediatric population followed in mental health outpatient and inpatient clinical settings: MEMAS prospective study protocol. BMJ Open. 2021 Jan 17;11(1):e040764. doi: 10.1136/bmjopen-2020-040764. PMID 33455928